CLINICAL TRIAL: NCT05414851
Title: Short-term Effects of a Low-carbohydrate Diet and a Whole-food, Plant-based Diet on Newer Markers of Vascular Health
Brief Title: Low-Carbohydrate and Plant-Based Dietary Effects on Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Thomas M Campbell, Assistant Professor of Family Medicine, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB 0007277
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Heart Disease, Ischemic; Hyperlipidemias; Hypertension
MeSH Terms: conditions — Myocardial Ischemia; Hyperlipidemias; Hypertension | interventions — Diet, Plant-Based; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: All subjects will consume two separate diets, with a 4-6 washout in between. They will be randomized 1:1 to determine which diet they start with.
Who Masked: Outcomes Assessor
Masking Description: Laboratory personnel will not know which dietary phase each subject has completed, but otherwise blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Food, Plant-Based Start (Experimental): This group starts with the whole-food, plant-based diet, then gets the low-carbohydrate diet after the washout period.
  Interventions: Other: Whole-Food, Plant-Based Diet and Low-Carbohydrate Diet
- Low-Carbohydrate Start (Experimental): This group starts with the low-carbohydrate diet, then gets the whole-food, plant-based diet after the washout period.
  Interventions: Other: Whole-Food, Plant-Based Diet and Low-Carbohydrate Diet

INTERVENTIONS:
Other: Whole-Food, Plant-Based Diet and Low-Carbohydrate Diet — Participants will consume two weeks of each diet, with a 4-6 week washout period in between. Meals and snacks are provided for convenience to enhance adherence to each dietary pattern, but subjects can add or include their own home-prepared foods as long as they meet dietary guidelines. Each dietary intervention will include an education session via Zoom teleconference, and at least 2 individual contacts by phone to address questions and assess for adverse events.

SUMMARY:
This is a randomized trial with a crossover design to investigate the short-term effects of two different dietary patterns on markers of vascular health. A low-carbohydrate diet and a whole-food, plant-based diet will be used. In addition to more traditional markers (cholesterol, blood pressure, inflammation), endothelial progenitor cells and trimethylamine N-oxide will be assessed.

DETAILED DESCRIPTION:
This study is an investigation of the short-term effects of two different diets on both conventional as well as newer markers of vascular health among subjects over the age of 50 who have a cardiovascular risk factor. The low-carbohydrate diet will be consistent with low-carbohydrate diet maintenance plans, with "net" carbs kept under 50g per day. The whole-food, plant-based diet will exclude animal foods, oils, and solid fats. Meals will be provided, and subjects will consume each diet for 2 weeks, with a 4-6 week washout period between dietary phases. Subjects will be randomized 1:1 to start with either the plant-based diet or the low-carbohydrate diet. Its primary aim is to assess the short-term effect of a whole-food, plant-based diet and a low-carbohydrate diet on levels of endothelial progenitor cells and trimethylamine N-oxide among this population. Secondarily, we will assess more conventional measures of vascular risk, including cholesterol, weight, blood pressure, insulin resistance, and inflammatory marker, as well as fullness and changes in nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

* Age >50
* Diagnosis of any of the following cardiovascular risk factors: hypertension (Diagnosis present in chart or use of antihypertensive medications); hyperlipidemia/dyslipidemia (non-HDL cholesterol ≥ 130 within the past year or current use of antihyperlipidemic medication); prediabetes (HbA1c ≥ 5.7% and < 6.5% in the past year); diabetes (HbA1c ≥ 6.5% in the past year); obesity (body mass index ≥ 30).
* Willing and able to comply with the protocol for the duration of the study, including food provision, scheduled meetings and testing visits.
* Able to speak and read English fluently because counseling and education is only available in English.

Exclusion Criteria:

* Active malabsorption syndrome (celiac disease, history of gastric bypass within the past year, uncontrolled Crohn's disease, protein-losing enteropathy, etc…)
* Use of any of the following medications that require close monitoring and adjustment during major dietary change: insulin, sulfonylureas, or warfarin
* Chronic or acute kidney disease, with eGFR < 50 on two or more lab tests in the past 6 months
* Diagnosis of cirrhosis or liver failure
* Hyperkalemia (defined as potassium >5.4 on two or more lab tests in the past 6 months)
* Major surgery in the past 3 months
* Myocardial infarction in the past 6 months
* Current, active eating disorder as determined by chart review, investigator assessment, or subject history
* Food allergies or intolerances that would interfere with eating study food or require special accommodation as determined by subject history, investigator assessment, or chart review
* Consuming a current diet described by the subject as vegetarian, vegan, very low-carbohydrate, or ketogenic
* Illicit drug use (not including marijuana)
* High risk alcohol use, based on subject history (defined as greater than 7 drinks/week for women and greater than 14 drinks/week for men)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Endothelial Progenitor Cells | 2 weeks
trimethylamine N-oxide | 2 weeks
HDL function | 2 weeks

SECONDARY OUTCOMES:
Cholesterol Panel | 2 weeks
  Total, LDL, HDL, non-HDL cholesterol, and triglycerides
Blood Pressure | 2 Weeks
Resting Heart Rate | 2 weeks
Weight | 2 weeks
Insulin resistance | 2 weeks
  HOMA-IR
Insulin | 2 weeks
Blood Glucose | 2 weeks
Inflammatory Markers | 2 weeks
  hsCRP, TNF-a, IL-6
Satiety Assessment | 2 weeks
  Adapted SLIM (satiety labeled intensity magnitude)
Food "liking" | 2 weeks
  5 food liking factor scales adapted from 5-Factor Satiety Questionnaires
Change in nutritional intake | 2 weeks
  assessed by 3 day food records at baseline and in second week of dietary phase

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Campbell, MD, Principal Investigator — University of Rochester
Locations (1):
- UR Medicine Nutrition in Medicine Research Center, Webster, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided